CLINICAL TRIAL: NCT07199751
Title: Vergleich Der Komplikationsrate, Des Funktionellen Outcomes Und Der Lebensqualität Zwischen Standard Therapie Versus Fast Track Therapie Bei Patienten Und Patientinnen Nach Hüft-TEP Operationen
Brief Title: Comparison of Complication Rate, Functional Outcome and Quality of Life Between Standard Therapy Versus Fast-track Therapy in Patients Following Hip Replacement Surgery
Status: Recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, BarbaraVogel, Dr. rer. biol. hum., Technical University of Munich
Other Study IDs: 2025-155-S-CB
Record Dates: First submitted 2025-07-07; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Coxarthrosis
Keywords: enhanced recovery; physiotherapy
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fast Track: enhanced Recovery
- standard therapy: standard therapy

SUMMARY:
The fast track group vs. control group will be compared with regard to hospitalization time and the non-inferiority of the fast track group vs. control group with regard to HOOS will be assessed.

The questionnaires will only be collected in the study: Eq-5d-5l, HOOS, self-efficacy, enjoyment of movement, fear of movement, pain catastrophizing.

DETAILED DESCRIPTION:
Around 400,000 hip and knee endoprostheses are implanted in Germany every year. Due to demographic change, the trend is clearly on the rise, which also results in rising costs in this area for the solidarity community. The Clinic for Orthopaedics and Sports Orthopaedics at the TUM Clinic is about to implement the Fast Track method after total hip arthroplasty (THA, in German: Hüft-TEP). The aim of this method is to shorten the length of stay in hospital and the post-operative recovery time as well as to promote rapid mobilization and independence of patients without worsening the functional outcome or the complication rate. The investigators will therefore investigate the extent to which it is possible to reduce the length of hospital stay without compromising function.

* Primary endpoints: Hospital length of stay, HOOS.
* Secondary endpoints: PROMs Quality of life Eq-5d-5l (EuroQol 5 dimensions Lang) Function Mobility (TUG test) in seconds Pain (NRS), ROM (neutral zero method), Strength (Nm/kg body weight, muscle function test) Self-efficacy/ pleasure/ fear of movement/pain catastrophizing Exercise self efficacy scale (ESES), physical activity enjoyment scale (PACES), Kinesiophobia (TSK), Pain catastrophizing scale (PCS).

With an original length of stay of 6 days and a target length of stay of 4 days, the expected reduction is 2 days. A standard deviation of 3 days is assumed in both groups (calculations based on patient data from August to December 2024) and a significance level of 0.05 and power of 80% are assumed. The required number of cases is therefore at least 36 participants per group. With this number of cases, the non-inferiority of the fast-track method compared to the standard method with regard to HOOS can also be demonstrated with a probability of 80%, assuming that the true mean difference between the methods is 0 points and the standard deviation for both methods is 15 points (Δ = 10 points, one-sided 97.5% confidence interval). To compensate for a potential drop-out rate, 45 patients per group should be recruited. With a primary hip TEP (THA) surgery rate of approx. 10 patients per week (cf. 2024) and a 2-month duration per group, the investigators can recruit a maximum of 80 patients per group. The investigators are therefore confident that the required case number of 45 per group will be reached.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* The patient will undergo surgery at Klinikum rechts der Isar, Technical University of Munich (TUM)
* Written informed consent for participation in the study after detailed explanation of the nature, significance, risks and scope of the clinical trial
* Written informed consent from the patient for data collection and data processing, with the patient fully informed.
* Sufficient German language skills of the patient.

Exclusion Criteria:

* Age < 18 years
* The patient is under guardianship, legally incapacitated or has limited legal capacity
* Only partial weight-bearing permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hip arthroplasty elective
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay (days) | From day of surgery until discharge, up to 4 days post-surgery
  The total number of days a participant remains admitted in the hospital from the day of surgery until discharge. While the expected length of stay is approximately 4 days, some participants may stay longer depending on clinical needs.
Hip Disability and Osteoarthritis Outcome Score (HOOS) | From baseline (pre-surgery) to 3 months post-surgery
  The Hip Disability and Osteoarthritis Outcome Score (HOOS) is a validated, patient-reported instrument for assessing hip-related pain, function, and quality of life.
  Scores range from 0 to 100, with higher scores indicating better outcomes (less pain, better function, improved quality of life).

SECONDARY OUTCOMES:
Timed Up and Go (TUG) Test | From baseline (pre-surgery) to 3 months post-surgery
  The Timed Up and Go (TUG) test is a functional mobility test measuring the time (in seconds) required for a participant to rise from a chair, walk 3 meters, turn, walk back, and sit down again. Shorter times indicate better functional mobility.
EQ-5D-5L (EuroQol 5 Dimensions, 5 Levels) | From baseline (pre-surgery) to 3 months post-surgery
  The EQ-5D-5L (EuroQol 5 Dimensions, 5 Levels) measures health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It also includes a visual analogue scale (VAS) for overall health.
  Index values are calculated using country-specific preference weights and typically range from 1 (full health) to 0 (equivalent to death), with negative values representing health states considered worse than death (e.g., -0.205 to 1.000 in Germany).
Range of Motion (ROM) - Neutral Zero Method (degrees) | From baseline (pre-surgery) to 3 months post-surgery
  Joint range of motion (ROM) assessed using the neutral zero method, measuring the maximal angle achieved at the hip joint. Higher values indicate greater mobility.
Exercise Self-Efficacy Scale (ESES) | From baseline (pre-surgery) to 3 months post-surgery
  The Exercise Self-Efficacy Scale (ESES) assesses an individual's confidence in their ability to engage in and maintain regular exercise, even under challenging circumstances, such as a busy work schedule, fatigue, being on vacation, or feeling stressed. Scores range from 6 to 60, with higher scores indicating greater self-efficacy for exercise.
Pain Catastrophizing Scale (PCS) | From baseline (pre-surgery) to 3 months post-surgery
  The Pain Catastrophizing Scale (PCS) measures the extent of negative thoughts and feelings related to pain.
  Scores range from 0 to 52, with higher scores indicating greater pain catastrophizing (worse outcome).
Tampa Scale for Kinesiophobia (TSK) | From baseline (pre-surgery) to 3 months post-surgery
  The Tampa Scale for Kinesiophobia (TSK) assesses fear of movement and avoidance of physical activity due to pain-related concerns.
  Scores range from 17 to 68, with higher scores indicating greater kinesiophobia (worse outcome).
Muscle Strength (Nm/kg body weight) | From baseline (pre-surgery) to 3 months post-surgery
  Maximal isometric muscle strength normalized to body weight, measured in Newton-meters per kilogram. Higher values indicate greater muscle strength.
Physical Activity Enjoyment Scale (PACES) | From baseline (pre-surgery) to 3 months post-surgery
  The Physical Activity Enjoyment Scale (PACES) assesses an individual's level of enjoyment during physical activity. Total scores range from 4 to 20, with higher scores indicating greater enjoyment of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Rüdiger von Eisenhart-Rothe, Prof. Dr., Study Director — Department of Orthopedics and Sports Orthopedics
Locations (1):
- Department Physical Therapy, München, Germany

IPD SHARING:
Plan to Share IPD: No